CLINICAL TRIAL: NCT05004519
Title: Impact of an Opioid Free Anesthesia Protocol Compared to Multimodal Anesthesia on Postoperative Morphine Consumption in an Enhanced Recovery After Gastric Bypass Surgery Protocol: a Prospective, Double Blind Study
Brief Title: Benefits of Opioid Free Anesthesia on Morphine Consumption in Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: matthieu clanet (Other)
Responsible Party: Sponsor-Investigator, matthieu clanet, Head of anesthesia department, Chirec
Organization: Chirec (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2021/378
Record Dates: First submitted 2021-08-03; First posted 2021-08-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Analgesics, Opioid
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid free anesthesia (Experimental): Dexmedetomidine 0,5 microgrammes/kg of ideal body weight (IBW) + magnesium 40 mg/kg of total body weight (TBW) in 10 minutes
  * Dexmedetomidine 0,4- 0,8 microgrammes/kg of IBW/h;Lidocaine 2% 49ml+ Ketamine 50mg: 1ml/10kg of IBW/ hour;Ketamine 25 mg;lidocaïne 1,5 mg/kg IBW;Propofol 2mg/kgTBW;Rocuronium 1,2 mg/kg IBW;Cefazoline 2g if >120 kg, 3g if >120Kg;Paracetamol 15 mg/ KgTBW;Diclofenac 75 mg;Dexamethasone 10 mg;Ondansetron 4 mg;Sevorane;dexmedetomidine: 0,4-0,8 microgramme/kg/h;Rocuronium 0,1 mg/kg of IBW if posttetanic count>1/10;Atropine 0,5 mg if heart rate < 40/min;Ephedrine 5mg in Arterial mean pressure < 20% of basal value;Nicardipine 0,5 mg if Arterial mean pressure > 20% of basal value Emergence
  * Stop dexmedetomidine;Stop sevorane;1 ml of NaCL 0,9%;Suggamadex 4 mg/ kg of IBW+ 4mg/kg of 40% ABW Post-anesthesia:Lidocaïne 2% 49ml + Ketamine 50 mg: 0,5 ml/ 10 kg IBW;Paracetamol 1g/6h;Diclofenac 75mg/12h;Morphine patient controlled analgesia: 1 mg/5 min, maximum 20mg/ 4 hours
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Multimodal anesthesia (Experimental): magnesium 40 mg/kg of total body weight (TBW) in 10 minutes
  * Remifentanil 0,2-0,4 microgrammes/kg/min of ideal body weight; Saline 0,9%: Infusion at 1ml/10kg of ideal body weight/ hour;Ketamine 25 mg;lidocaïne 1,5 mg/kg IBW;Propofol 2mg/kgTBW;Rocuronium 1,2 mg/kg IBW;Cefazoline 2g if >120 kg, 3g if >120Kg;Paracetamol 15 mg/ Kg TBW;Diclofenac 75 mg;Dexamethasone 10 mg;Ondansetron 4 mg;Sevorane;remifentanil 0,2-0,4 microgrammes/kg/min;Rocuronium 0,1 mg/kg of IBW if posttetanic count>1/10;Atropine 0,5 mg if heart rate < 40/min;Ephedrine 5mg in Arterial mean pressure < 20% of basal value;Nicardipine 0,5 mg if Arterial mean pressure > 20% of basal value Emergence
  * Stop remifentanil;Stop sevorane;1 ml of morphine 10mg/ml;Suggamadex 4 mg/ kg of IBW+ 4mg/kg of 40% ABW Post-anesthesia:Salne 50ml: 0,5 ml/ 10 kg IBW;Paracetamol 1g/6h;Diclofenac 75mg/12h;Morphine patient controlled analgesia: 1 mg/5 min, maximum 20mg/ 4 hours
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — dexmedetomidine or remifentanil during laparoscopic gastric bypass
  Arms: Opioid free anesthesia
Drug: Remifentanil — dexmedetomidine or remifentanil during laparoscopic gastric bypass
  Arms: Multimodal anesthesia

SUMMARY:
Opioid free anesthesia is a recent anesthesia technique with the aim to avoid peroperative use of morphinics to allow a diminution of secondary morphinics effects in the postoperative period.

There is no robust data on the real benefits of such procedures. Obese patients are particular at risk of secondary effects of opioids. The aim of our study is to compare opioid free anesthesia to multimodal anesthesia on postoperative morphine consumption after a laparoscopic gastric bypass.

DETAILED DESCRIPTION:
The aim of the study is to study the impact of an opioid free anesthesia protocol on the postoperative morphine consumption in laparoscopic gastric bypass compared to a multimodal anesthesia protocol.

183 morbidly obese patients (Body mass index >40Kg/m2 or >35kg/m2 AND/OR diabete mellitus AND/OR sleep apnea syndrome AND/OR arterial hypertension.

A randomization will allocate two groups of 100 patients in:

* Group 1: Multimodal anesthesia without opioids
* Group 2: Multimodal anesthesia with opioid The patient, the anesthesist and the data evaluator will be all blinded about the allocation of the patient.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anesthesia score (ASA) 2-3
* Scheduled for a laparoscopic gastric bypass surgery

Exclusion Criteria:

* Patient refusal
* Medical diseases: Cardiac arrhythmia like atrioventricular block 2nd or 3rd degree, pacemaker, arterial hypotension, severe bradycardia, cerebrovascular pathology, renal and/or hepatic insufficiency
* Previous bariatric surgery
* Allergy to any medication used during the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Total Morphine consumption | 24 hours after surgery
  total morphine consumption from the PACU arrival to the 24 h post-surgery

SECONDARY OUTCOMES:
Visual analog scale | Post Anesthesia Care Unit admission (Hour 0), Hour +4, Hour +24
Morphine consumption | Post Anesthesia Care Unit admission (Hour 0), Hour +4
Quality of Recovery 40 score | operative Day -1, Operative day +1, operative day +30
  Recovery scale: From 40 (worst recovery) to 200 (Best Recovery)
Hypoxemia | up to patient discharge
  SpO2 < 90% on 2 liters of nasal Oxygen
Postoperative Nausea and vomiting | Post Anesthesia Care Unit admission (Hour 0), Hour +4, Hour +24
Need of Antiemetics | Up to patient discharge
Bradycardia and use of atropine | Up to patient discharge
Readmissions rate | Up to 30 days
  Admission of the patient in hospital during the first 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: matthieu Clanet, Principal Investigator — Chirec
Locations (1):
- CHIREC Delta Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Study protocol, informed consent form

REFERENCES:
- [Derived] Clanet M, Touihri K, El Haddad C, Goldsztejn N, Himpens J, Fils JF, Gricourt Y, Van der Linden P, Coeckelenbergh S, Joosten A, Dandrifosse AC. Effect of opioid-free versus opioid-based strategies during multimodal anaesthesia on postoperative morphine consumption after bariatric surgery: a randomised double-blind clinical trial. BJA Open. 2024 Feb 23;9:100263. doi: 10.1016/j.bjao.2024.100263. eCollection 2024 Mar. PMID 38435809